CLINICAL TRIAL: NCT01518621
Title: Whole Brain Radiation With or Without Erlotinib for Brain Metastases From Non-Small Cell Lung Cancer
Acronym: RadEr
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: Oslo University Hospital (Other)
Responsible Party: Principal Investigator, Odd Terje Brustugun, Senior consultant, Oslo University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RadEr
Record Dates: First submitted 2012-01-19; First posted 2012-01-26 (Estimated); Last update posted 2019-03-13 (Actual); Status verified 2019-03

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms | interventions — Radiation; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Radiotherapy alone (Active Comparator): Total brain irradiation, 3Gy x10
  Interventions: Radiation: Radiation
- Radiation plus erlotinib (Experimental): Total brain irradiation, 3Gy x10 plus erlotinib 150 mg q d from radiation day -1 through last day of irradiation
  Interventions: Drug: Radiation plus erlotinib

INTERVENTIONS:
Radiation: Radiation — Whole brain radiation
  Other Names: Whole brain radiation therapy
  Arms: Radiotherapy alone
Drug: Radiation plus erlotinib — Radiation 3Gy x10 plus erlotinib 150 mg q d, from the day before radiation start, through last day of irradiation
  Other Names: Whole brain radiation therapy and tyrosin kinase inhibitor
  Arms: Radiation plus erlotinib

SUMMARY:
To determine if erlotinib given orally along with concurrent whole brain irradiation in lung cancer patients with brain metastases improves median overall survival and enhances local control compared to those treated with WBRT alone, without significantly increasing the risk of side effects or lowering quality of life.

DETAILED DESCRIPTION:
Endpoints

Primary:

• To determine if erlotinib given orally along with concurrent WBRT in lung cancer patients with brain metastases, improves median overall survival compared to those treated with WBRT alone.

Secondary:

* To confirm the safety profile of erlotinib along with concurrent WBRT, in the context of treating central nervous system malignancies.
* To evaluate if erlotinib along with concurrent WBRT increases local control rate as measured by MRI at 8 weeks, compared to WBRT alone.
* To evaluate if erlotinib along with concurrent WBRT increases time to neurologic progression of disease based on neuropsychological assessment at baseline, at 8 and 20 weeks after WBRT.
* To evaluate quality of life parameters in patients treated with WBRT alone vs concomitant erlotinib and WBRT
* To evaluate if mutation status has impact on the above mentioned parameters Trial design Open multicenter randomized phase II trial. Patients Patients > 18 years with histologically confirmed NSCLC and brain metastases verified on either CT or MRI, not eligible for neurosurgery or stereotactic radiation therapy.

Trial treatment Patients will be randomized 1:1 to either treatment arm A or B.

* Arm A: WBRT 3 Gy x10 alone.
* Arm B: WBRT 3 Gy x10 and erlotinib given concomitantly, 150 mg p.o. daily from the day before radiation, until the last day of radiation.

Number of patients 150 patients will be included, 75 in each arm

ELIGIBILITY:
Inclusion Criteria: Histologically or cytologically confirmed advanced non-small cell lung cancer (NSCLC) meeting 1 of the following criteria:

* Newly diagnosed multiple brain metastases not suitable for first-line chemotherapy
* Relapsed NSCLC with newly diagnosed multiple brain metastases
* Relapsed NSCLC after second-line or more chemotherapy regimens with newly diagnosed multiple brain metastases

  * Diagnosis of brain metastases confirmed by MRI (or CT if MRI is not available/possible) within the past 4 weeks
  * Symptoms attributable to brain metastases
  * Patients who have undergone craniotomy with incomplete resection are eligible
  * Clinician's opinion that whole-brain radiotherapy (WBRT) will be beneficial
  * ECOG PS 0-2
  * Age above 18 years
  * Serum bilirubin < 2 times upper limit of normal (ULN)
  * AST and ALT < 2 times ULN (< 5 times ULN if liver metastases are present)
  * Creatinine < 1.5 times ULN
  * Able to take oral medication
  * Not pregnant or nursing
  * Negative pregnancy test
  * Fertile patients must use effective contraception
  * No other prior or concurrent malignant disease likely to interfere with study treatment or comparisons

Exclusion Criteria:

* More than 3 sites (organ systems) of extracranial metastases
* Evidence of solitary brain metastasis on MRI that can be treated with surgical resection, radiosurgery, or stereotactic radiotherapy
* Evidence of other significant laboratory finding or concurrent uncontrolled medical illness, that in the opinion of the investigator, would interfere with study treatment or results comparison or render the patient at high risk for treatment complications

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2012-05; Primary Completion 2017-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Odd Terje Brustugun, MD PhD, Principal Investigator — Norwegian Radium Hospital
Locations (1):
- The Norwegian Radium Hospital, Oslo, Norway